CLINICAL TRIAL: NCT00181038
Title: Analgesia of Fibula Free Flap Donor Site by Peri-Neuronal Catheter in Oro-Pharyngeal Carcinoma Surgery: Comparing Continuous Infusion of Local Anesthetic With Systemic Multimodal Analgesia
Brief Title: Analgesia of Fibula Free Flap Donor Site by Peri-Neuronal Catheter in Oro-Pharyngeal Carcinoma Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PERONE; CSET 2003/1042
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-08-28 (Estimated); Status verified 2006-09

CONDITIONS: Oropharyngeal Neoplasms
Keywords: Oro-Pharyngeal Carcinoma Surgery
MeSH Terms: conditions — Oropharyngeal Neoplasms

INTERVENTIONS:
Device: Peri-Neuronal Catheter

SUMMARY:
This trial examines the analgesia of the fibula free flap donor site by peri-neuronal catheter in oro-pharyngeal carcinoma surgery by comparing continuous infusion of a local anesthetic with systemic multimodal analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for oro-pharyngeal carcinoma surgery with reconstruction by fibula free flap

Exclusion Criteria:

* Allergy to propofol or local anesthetic (ropivacaine)
* Severe renal or cardiac failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-06

PRIMARY OUTCOMES:
Assess the influence of locoregional anesthesia on postoperative morphine consumption

SECONDARY OUTCOMES:
Visual analog pain scale on the free flap donor site

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Plantevin, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France